CLINICAL TRIAL: NCT00352638
Title: Colorectal Cancer Screening Intervention for Family Members of Colorectal Cancer Patients
Brief Title: Educational Intervention With or Without Telephone Counseling in Increasing Colorectal Cancer Screening Compliance in Brothers and Sisters of Patients With Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized
Other Study IDs: FCCC-FCRB-04-004-P; CDR0000485294 (Registry Identifier: PDQ (Physician Data Query)); FCCC-00-841; NCT00491205 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention
Other: educational intervention
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Printed educational materials and counseling by telephone may improve colorectal cancer screening compliance in brothers and sisters of patients with colorectal cancer.

PURPOSE: This randomized phase III trial is studying standard or personalized printed educational materials with or without telephone counseling to compare how well they work in increasing colorectal cancer screening compliance in brothers and sisters of patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the impact of 3 interventions (generic educational print intervention, tailored educational print intervention, or tailored educational print intervention plus telephone counseling) on colorectal cancer screening behaviors and intentions among siblings at increased familial risk for colorectal cancer.

Secondary

* Determine whether demographic factors, medical access, physician recommendation at baseline, and proband (patient) characteristics (e.g., stage of disease) moderate the impact of the interventions on colorectal screening.
* Evaluate whether knowledge, attitude, and physician recommendation variables mediate the association between the interventions and colorectal screening, and determine whether these variables are impacted by the interventions.
* Analyze the cost of each intervention.

OUTLINE: This is a randomized, controlled, cohort, multicenter study. Participants are stratified according to study site. Participants are randomized to 1 of 3 intervention arms.

* Arm I: Participants receive generic educational print intervention approximately 1 week after completing the baseline survey.
* Arm II: Participants receive tailored educational print intervention within 10 days after completing the baseline survey and a tailored newsletter 1 month after completing the baseline survey.
* Arm III: Participants receive tailored educational print intervention approximately 14-18 days after completing the baseline survey. Participants undergo a telephone counseling session within 2 weeks after receiving the tailored print intervention and receive a tailored newsletter 1 month after completing the baseline survey.

After study completion, participants are followed at 6 months and/or 1 year.

PROJECTED ACCRUAL: A total of 660 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Sibling of a patient diagnosed with adenocarcinoma of the colon or rectum

  * Patient (proband) must meet the following criteria:

    * Diagnosed in 1999 or later
    * Currently living
    * Seen in Community Clinical Oncology Program member hospital
    * 60 and under at diagnosis
* No history of hereditary cancer syndrome (e.g., familial adenomatous polyposis or hereditary nonpolyposis colorectal cancer) (patient and sibling)
* No history of colorectal cancer or colorectal polyps (sibling)
* No history of inflammatory bowel disease (patient and sibling)

PATIENT CHARACTERISTICS:

* Age 40 and over OR within 10 years of proband's (patient's) age at diagnosis
* English speaking

PRIOR CONCURRENT THERAPY:

* No prior colorectal cancer screening

  * May have undergone prior screening provided they have not followed, or do not plan to follow, physician's recommendation for screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2005-08; Primary Completion 2012-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening compliance

SECONDARY OUTCOMES:
Impact on movement in stage of adoption
Increased knowledge and attitudes
Cost

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (18):
- United States (18):
  - Helen F. Graham Cancer Center at Christiana Care, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center CCOP Research Base, Tampa, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Northeast Regional Cancer Institute, Scranton, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas